CLINICAL TRIAL: NCT04280133
Title: A Randomized Controlled Trial of an Educational Video Tool for Patients Receiving CAR T-Cell Therapy
Brief Title: CAR T-CELL Therapy Educational Video Trial
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Patrick C. Johnson, MD, Principal Investigator, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 19-790
Record Dates: First submitted 2020-02-19; First posted 2020-02-21 (Actual); Last update posted 2023-01-26 (Actual); Status verified 2023-01

CONDITIONS: Hematologic Malignancy; CAR-T Cell Therapy
Keywords: Hematologic Malignancy; CAR-T cell therapy
MeSH Terms: conditions — Hematologic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Educational Video Tool (Experimental): Patients randomized to the intervention arm will watch a 3-minute video educational tool about CAR-T cell therapy prior to admission for CAR-T cell therapy.
  Interventions: Behavioral: Educational Video Tool
- Standard Care (No Intervention): Patients randomized to the control arm will receive usual care per the treating team. Any questions regarding CAR-T cell therapy will be directed to the patient's medical team

INTERVENTIONS:
Behavioral: Educational Video Tool — The video educational tool was written by the investigators in collaboration with a panel of experts on CAR T-cell therapy, medical ethicists, palliative care clinicians, and oncologists.
  Arms: Educational Video Tool

SUMMARY:
The purpose of this study is to test a new educational video to help patients and doctors talk about CAR-T cell therapy, a treatment being used in cancer.

- Educational video tool for patients receiving CAR-T cell therapy.

DETAILED DESCRIPTION:
This research study is a Feasibility Study, which is the first-time investigators are examining this educational video tool for patients receiving CAR-T cell therapy.

The research study procedures include screening for eligibility, randomization and a series of questionnaires

Participants will be randomized to one of 2 groups:

* Group A: Educational video tool
* Group B: Standard care

Participants will be in the research study for a month after consent

It is expected that about 80 participants will take part in this research study.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or age or older
* Established diagnosis of a hematologic malignancy
* Under consideration for CAR T-cell therapy at Massachusetts General Hospital

Exclusion Criteria:

* Significant uncontrolled psychiatric disorders (psychotic disorder, bipolar disorder, major depression) or other co-morbid disease (dementia, cognitive impairment), which the primary oncologist believes prohibits informed consent or participation in the study
* Undergoing CAR T-cell therapy for solid tumor malignancy
* Inability to comprehend English, as the video is currently only available in English at this time

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2020-05-25 (Actual); Primary Completion 2022-10-26 (Actual); Study Completion 2023-02-24 (Estimated)

PRIMARY OUTCOMES:
Feasibility (enrollment and retention rates) | Up to 1 year
  The primary endpoint is feasibility. The proposed video intervention will be deemed feasible if at least 60% of eligible patients are enrolled in the study.

SECONDARY OUTCOMES:
Knowledge about CAR-T cell therapy (CAR-T cell Knowledge Questionnaire) | up to 1 month
  To compare patient's knowledge about CAR-T cell therapy between groups as measured by the CAR-T cell therapy Knowledge Questionnaire (Score range 0-10). Higher scores indicating higher knowledge.
Psychological distress (Hospital Anxiety and Depression Scale (HADS) | up to 1 month
  To compare patient's psychological distress between groups as measured by the HADS. HADS Anxiety and Depression subscales range from 0-21, with higher scores indicating worse psychological distress.
Patient's self-efficacy (modified version of CASE-cancer) | up to 1 month
  To compare patient's self-efficacy between the groups as measured by a modified version of the Communication and Attitudinal Self-Efficacy Scale-Cancer (CASE-cancer) for patients receiving CAR-T cell therapy. The modified CASE ranges from 0-170 with higher scores indicating higher self-efficacy
Preferences for CAR T-cell therapy (single-item preference for CAR-T cell therapy) | up to 1 week
  To compare patient's preferences for CAR-T cell therapy between groups as measured by a single-item "Do you prefer to receive CAR-T cell therapy". We will compare proportion of patients stating "yes" to receiving CAR-T cell therapy between groups.
Decision Satisfaction around receipt of CAR-T cell therapy | up to 1 month
  To compare patient's satisfaction around the decision to receive CAR-T cell therapy between groups as measured by a five-item Likert scale ranging from "Strongly Disagree" to "Strongly Agree" with statements about satisfaction regarding the decision to receive CAR-T cell therapy, with "Strongly Agree" indicating the highest decision satisfaction. We will compare the proportion of patients stating "Agree" or "Strongly Agree" to the six items between groups.
Acceptability of the video (intervention arm only) | up to 1 month
  To assess, in the intervention group only, patients' comfort with watching the video, whether they find the video helpful in their understanding of CAR T-cell therapy, and whether they would recommend it to others as measured by a 3-item survey. Each of the three items is a four-point Likert scale. Acceptability is defined as at least 80% of patients intervention reporting they felt "very comfortable" or "somewhat comfortable" on a four-point Likert scale when asked about their comfort watching the video.

CONTACTS AND LOCATIONS:
Overall Officials: Patrick C Johnson, MD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
The Dana-Farber / Harvard Cancer Center encourages and supports the responsible and ethical sharing of data from clinical trials. De-identified participant data from the final research dataset used in the published manuscript may only be shared under the terms of a Data Use Agreement. Requests may be directed to Sponsor Investigator or designee. The protocol and statistical analysis plan will be made available on Clinicaltrials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data can be shared no earlier than 1 year following the date of publication
Access Criteria: Contact the Partners Innovations team at http://www.partners.org/innovation